CLINICAL TRIAL: NCT05896449
Title: Predictive Values of Preoperative [68Ga]Ga-PSMA-11 PET/CT in Patients With Suspected Brain Tumours of Glial Origin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WUM-ZMN-05-2023
Record Dates: First submitted 2023-05-17; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Glioma, Malignant; Glioma Glioblastoma Multiforme
Keywords: glioma; PSMA; PET/CT; [68Ga]Ga-PSMA-11 PET/CT; glial tumours
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/CT before surgery (Experimental): [68Ga]Ga-PSMA-11 PET/CT before surgery
  Interventions: Diagnostic Test: [68Ga]Ga-PSMA-11 PET/CT

INTERVENTIONS:
Diagnostic Test: [68Ga]Ga-PSMA-11 PET/CT — The PET/CT image acquisition was performed from the skull to the mid-thigh (3-min per bed position, 3 iterations, 21 subsets) with a CT scan (120 kV, 170mAs reference) with dose modulation for anatomic correlation (CARE dose 4D) and attenuation correction on a Biograph 64 TruePoint (Siemens Medical Solutions Inc., USA) 60 min post injection of [68Ga]Ga-PSMA-11 (2 MBq per kg body weight).

SUMMARY:
The aim of this study was to analyse usefulness of [68Ga]Ga-PSMA-11 PET/CT scans in preoperative differentiation between HGG and LGG in patients with suspicion of a tumor of glial origin in previously performed imaging examinations. The PET/CT scan will be compared with postoperative histopathological results and with additional immunohistochemical staining for PSMA expression.

ELIGIBILITY:
Inclusion Criteria:

* primary lesion found in CT/MRI with radiological features of glial neoplasm
* untreated disease, planned surgery
* negative medical history of other neoplastic diseases
* age over 18
* informed, voluntary consent to participate in the study

Exclusion Criteria:

* pregnant women, breastfeeding women
* persons with a known allergy to PSMA
* age under 18
* patient's lack of cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
PET/CT vs histopathological diagnosis | through study completion, an average of 1.5 year
  Comparison of the incidence of positive preoperative [68Ga]Ga-PSMA-11 PET/CT results with the final histopathological diagnosis based on the 5th edition of the WHO (World Health Organization) Classification of Tumours of the Central Nervous System (2021).
  The PET scan in this regard will be evaluated qualitatively - in terms of finding accumulation in the projection of the brain tumor (positive result) and lack of accumulation in the projection of the brain tumor (negative result).
  The histopathological diagnosis will take into account the subtypes of the tumor according on the 5th edition of the WHO (World Health Organization) Classification of Tumours of the Central Nervous System (2021) - including the histopathological examination and the genetic diagnosis - adult-type diffuse gliomas comprise of three distinct types: Astrocytoma, IDH-mutant, Oligodendroglioma, IDH-mutant and 1p/19q-codeleted, and Glioblastoma, IDH-wildtype

SECONDARY OUTCOMES:
PET/CT semiquantitive parameter - SUVmax vs histopathological diagnosis | through study completion, an average of 1.5 year
  Comparison of the preoperative [68Ga]Ga-PSMA-11 PET/CT semiquantitative parameters with with the final histopathological diagnosis.
  The maximal standard uptake value (SUVmax) of each positive lesion were measured using the spherical volume of interest (VOI).
  The histopathological diagnosis will take into account the subtypes of the tumor according on the 5th edition of the WHO (World Health Organization) Classification of Tumours of the Central Nervous System (2021) - including the histopathological examination and the genetic diagnosis - adult-type diffuse gliomas comprise of three distinct types: Astrocytoma, IDH-mutant, Oligodendroglioma, IDH-mutant and 1p/19q-codeleted, and Glioblastoma, IDH-wildtype.
PET/CT semiquantitive parameter SUVmean vs histopathological diagnosis | through study completion, an average of 1.5 year
  Comparison of the preoperative [68Ga]Ga-PSMA-11 PET/CT semiquantitative parameters with with the final histopathological diagnosis.
  The mean standard uptake value (SUVmean) of each positive lesion were measured using the spherical volume of interest (VOI).
  The histopathological diagnosis will take into account the subtypes of the tumor according on the 5th edition of the WHO (World Health Organization) Classification of Tumours of the Central Nervous System (2021) - including the histopathological examination and the genetic diagnosis - adult-type diffuse gliomas comprise of three distinct types: Astrocytoma, IDH-mutant, Oligodendroglioma, IDH-mutant and 1p/19q-codeleted, and Glioblastoma, IDH-wildtype.
PET/CT semiquantitive parameter - TBR vs histopathological diagnosis | through study completion, an average of 1.5 year
  Comparison of the preoperative [68Ga]Ga-PSMA-11 PET/CT semiquantitative parameters with with the final histopathological diagnosis.
  The Target-to-background ratios (TBR) were calculated using SUVmax of the lesion divided by SUVmax of the background measured using a VOI of a similar diameter, placed in a distant, unaffected region, representing normal brain tissue.
  The histopathological diagnosis will take into account the subtypes of the tumor according on the 5th edition of the WHO (World Health Organization) Classification of Tumours of the Central Nervous System (2021) - including the histopathological examination and the genetic diagnosis - adult-type diffuse gliomas comprise of three distinct types: Astrocytoma, IDH-mutant, Oligodendroglioma, IDH-mutant and 1p/19q-codeleted, and Glioblastoma, IDH-wildtype.
PET/CT semiquantitive parameter - TLR vs histopathological diagnosis | through study completion, an average of 1.5 year
  Comparison of the preoperative [68Ga]Ga-PSMA-11 PET/CT semiquantitative parameters with with the final histopathological diagnosis.
  Target-to-liver background ratios (TLR) were calculated by dividing SUVmax of the lesion by SUVmean of the liver (the liver VOI of a similar diameter placed in the central area of the right liver lobe was used).
  The histopathological diagnosis will take into account the subtypes of the tumor according on the 5th edition of the WHO (World Health Organization) Classification of Tumours of the Central Nervous System (2021) - including the histopathological examination and the genetic diagnosis - adult-type diffuse gliomas comprise of three distinct types: Astrocytoma, IDH-mutant, Oligodendroglioma, IDH-mutant and 1p/19q-codeleted, and Glioblastoma, IDH-wildtype.
PET/CT semiquantitive parameter - SUVmax vs immunohistopathological staining | through study completion, an average of 1.5 year
  Comparison of the preoperative [68Ga]Ga-PSMA-11 PET/CT with the immunohistopathological staining of the tumour tissue.
  The maximal standard uptake value (SUVmax) of each positive lesion were measured using the spherical volume of interest (VOI).
  The immunoreaction will be analyzed in the endothelium and in tumor cells. A score will be assigned semiquantitatively based on staining intensity and distribution as follows: 0 - negative, 1- faint and weak staining at high power; 2- moderate intensity at low power; and 3- strong reaction at low power.
PET/CT vs progession free survival time. | 1 year after the study
  Comparison of the incidence of positive preoperative [68Ga]Ga-PSMA-11 PET/CT results with the progession free survival time.
  The PET scan in this regard will be evaluated qualitatively - in terms of finding accumulation in the projection of the brain tumor (positive result) and lack of accumulation in the projection of the brain tumor (negative result).
  The time will be measured in weeks.
PET/CT vs overall survival time. | 1 year after the study
  Comparison of the incidence of positive preoperative [68Ga]Ga-PSMA-11 PET/CT results with the overall survival time.
  The PET scan in this regard will be evaluated qualitatively - in terms of finding accumulation in the projection of the brain tumor (positive result) and lack of accumulation in the projection of the brain tumor (negative result).
  The time will be measured in weeks.
PET/CT semiquantitive parameter - SUVmax vs progession free survival time. | 1 year after the study
  Comparison of the incidence of positive preoperative [68Ga]Ga-PSMA-11 PET/CT results with progession free survival time.
  The maximal standard uptake value (SUVmax) of each positive lesion were measured using the spherical volume of interest (VOI).
  The time will be measured in weeks.
PET/CT semiquantitive parameter - SUVmax vs overall survival time. | 1 year after the study
  Comparison of the incidence of positive preoperative [68Ga]Ga-PSMA-11 PET/CT results with the overall survival time.
  The maximal standard uptake value (SUVmax) of each positive lesion were measured using the spherical volume of interest (VOI).
  The time will be measured in weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear Medicne Department Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 5 years
Access Criteria: reasoned request

REFERENCES:
- [Derived] Pelka K, Koczyk K, Koperski L, Dziedzic T, Nowak A, Krolicki L, Kunert P, Kunikowska J. Imply on diagnosis and early prognosis of preoperative [68Ga]Ga-PSMA-11 PET/CT in patients with suspected brain tumours of glial origin. Sci Rep. 2025 Jan 2;15(1):214. doi: 10.1038/s41598-024-84036-5. PMID 39747932